CLINICAL TRIAL: NCT02204033
Title: A Phase I Dose Escalation Study With 99mTC - or 186 Re-labelled Humanised Monoclonal Antibody BIWA 4, in Patients With Head and Neck Cancer
Brief Title: Dose Escalation Study With 99mTC - or 186 Re-labelled Humanised Monoclonal Antibody (hMAb) BIWA 4 in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1170.1
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

ARMS (4):
- 99mTc - labelled hMAb BIWA 4 - low dose (Experimental)
  Interventions: Drug: 99mTc - labelled hMAb BIWA 4; Drug: unlabelled hMAb BIWA 4 - low dose
- 99mTc - labelled hMAb BIWA 4 - medium dose (Experimental)
  Interventions: Drug: 99mTc - labelled hMAb BIWA 4; Drug: unlabelled hMAb BIWA 4 - medium dose
- 99mTc - labelled hMAb BIWA 4 - high dose (Experimental)
  Interventions: Drug: 99mTc - labelled hMAb BIWA 4; Drug: unlabelled hMAb BIWA 4 - high dose
- 186 Re - labelled hMAb BIWA 4 - escalating dose (Experimental)
  Interventions: Drug: 186 Re - labelled hMAb BIWA 4

INTERVENTIONS:
Drug: 99mTc - labelled hMAb BIWA 4
  Arms: 99mTc - labelled hMAb BIWA 4 - high dose; 99mTc - labelled hMAb BIWA 4 - low dose; 99mTc - labelled hMAb BIWA 4 - medium dose
Drug: 186 Re - labelled hMAb BIWA 4
  Arms: 186 Re - labelled hMAb BIWA 4 - escalating dose
Drug: unlabelled hMAb BIWA 4 - low dose
  Arms: 99mTc - labelled hMAb BIWA 4 - low dose
Drug: unlabelled hMAb BIWA 4 - medium dose
  Arms: 99mTc - labelled hMAb BIWA 4 - medium dose
Drug: unlabelled hMAb BIWA 4 - high dose
  Arms: 99mTc - labelled hMAb BIWA 4 - high dose

SUMMARY:
The general aim of the present study was to assess the safety and tolerability of intravenously administered Technetium 99m (99mTc) and Rhenium-186 radionuclide (186 Re) -labelled hMAb BIWA 4, to confirm preferential accumulation in the tumour of 99mTc - labelled hMAb BIWA 4, to determine the maximum tolerated radiation dose of 186 Re-labelled hMAb BIWA 4 and to propose a safety dose for phase II development.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmation of squamous cell carcinoma in the head and neck
* Patients destined for surgery by means of neck dissection (Part A) or :
* Patients with either local and/or regional recurrent disease for which curative treatment options were not available or distant metastases. The tumor deposits had to be measurable either clinically or by one or more radiological technique (s) (CT, MRI, bone scintigraphy). Because RIT was expected to be more effective in smaller size tumor deposits, patients with lesions measuring > 3 cm in greatest dimension were preferred (Part B)
* Patients over 18 years of age
* Patients younger than 80 years of age
* Patients who had given 'written informed consent'
* Patients with a life expectancy of at least 3 months
* Patients with a good performance status: Karnofsky > 60

Exclusion Criteria:

* Life-threatening infection, allergic diathesis, organ failure (bilirubin > 30µmol/l and/or creatinine > 150 µmol/l) or evidence of a recent myocardial infarction on ECG or unstable angina pectoris
* Pre-menopausal women (last menstruation <= 1 year prior to study start)

  * Not surgically sterile (hysterectomy, tubal ligation) and
  * Not practicing acceptable means of birth control, (nor not planned to be continued throughout the study). Acceptable methods of birth control include oral, implantable or injectable contraceptives
* Women with a positive serum pregnancy test at baseline
* Chemotherapy or radiotherapy within 4 weeks before inclusion in the study
* White blood cell count < 3000/mm³, granulocyte count < 1500/mm³ or platelet count < 100000/mm³
* Hematological disorders, congestive heart failure, bronchial asthma, alimentary or contact allergy, severe atopy or allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1999-03; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 10 weeks
Presence of human-anti-human-antibody (HAHA) | after 144 hours post infusion
Number of patients with clinically significant changes in vital signs | up to 6 weeks after infusion
Biodistribution of 99mTC-labelled hMAb BIWA 4 in tumour and normal tissue samples - Biopsy (Part A) | at 48 h after infusion
  uptake expressed as percentage of the injected dose per kg tissue (%ID/kg)
Immunoscintigraphic imaging evaluation (Parts A + B) | up to 21 hours after infusion
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 336 hours after infusion
Cmax (Maximum measured concentration of the analyte in plasma) | up to 336 hours after infusion
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 336 hours after infusion
t½ (Terminal half-life of the analyte in plasma) | up to 336 hours after infusion
Vz (Apparent volume of distribution during the terminal phase) | up to 336 hours after infusion
Vss (Apparent volume of distribution under steady-state conditions) | up to 336 hours after infusion
CL (Total body clearance) | up to 336 hours after infusion
MRT (Mean residence time) | up to 336 hours after infusion
Cumulative urinary excretion of radioactivity over time | up to 96 hours after infusion
Number of patients with abnormal changes in laboratory parameters | up to 6 weeks after infusion
Occurence of dose limiting toxicities (DLT) | up to 144 hours post infusion
Uptake of 99mTC-labelled hMAb BIWA 4 in tumour and normal tissue samples (Part A) | up to 6 weeks after infusion
  Assessment of biodistribution by radioimmunoscintigraphy expressed as low, medium or high
Actual organ uptake of 99mTC-labelled hMAb BIWA 4 | at 21 h after infusion
  expressed as % I.D. (injected dose)

SECONDARY OUTCOMES:
Tumour response according to response criteria of the World Health Organisation (WHO) | up to 144 hours after infusion
  assessed by Computer Tomography (CT) and/or by Magnet resonance imaging (MRI) and/or bone scintigraphy and/or by physical examination
Maximum tolerated radiation dose of 186Re-labelled hMAb BIWA 4 | up to 144 hours after infusion